CLINICAL TRIAL: NCT01167374
Title: Phase I Study Evaluating the Treatment of Patients With Hepatocellular Carcinoma (HCC) With Carbon Ion Radiotherapy
Brief Title: Carbon Ion Radiotherapy for Hepatocellular Carcinoma
Acronym: PROMETHEUS-01
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMETHEUS-01
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbon Ion Radiotherapy (Experimental): Increasing Dose of Carbon Ion Radiotherapy 4 x 10 Gy E to 4 x 14 Gy E
  Interventions: Radiation: Carbon Ion Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Increasing Dose of Carbon Ion Radiotherapy 4 x 10 Gy E to 4 x 14 Gy E

SUMMARY:
Treatment options for patients with advanced hepatocellular carcinoma (HCC) are often limited. In most cases, they are not amenable to local therapies including surgery or radiofrequency ablation. The multi-kinase inhibitor sorafenib has shown to increase overall survival in this patient group for about 3 months.

Radiation therapy is a treatment alternative, however, high local doses are required for long-term local control. However, due to the relatively low radiation tolerance of liver normal tissue, even using stereotactic techniques, delivery of sufficient doses for successful local tumor control has not be achieved to date.

Carbon ions offer physical and biological characteristics. Due to their inverted dose profile and the high local dose deposition within the Bragg peak precise dose application and sparing of normal tissue is possible. Moreover, in comparison to photons, carbon ions offer an increased relative biological effectiveness (RBE), which can be calculated between 2 and 3 depending on the HCC cell line as well as the endpoint analyzed.

Japanese Data on the evaluation of carbon ion radiation therapy showed promising results for patients with HCC.

In the current Phase I-PROMETHEUS-01-Study, carbon ion radiotherapy will be evaluated for patients with advanced HCC. The study will be performed as a dose-escalation study evaluating the optimal carbon ion dose with respect to toxicity and tumor control.

Primary endpoint is toxicity, secondary endpoint is progression-free survival and response.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed HCC or diagnosis of HCC according to AASLD-guidelines
* macroscopic tumor
* liver-confined disease without extrahepatic disease as diagnosed by CT, MRT, ultrasound and bone scan
* minimal distance of tumor edge to the intestines of 1cm
* age ≥ 18 years of age
* Karnofsky Performance Score ³60
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy of the hepatobiliary system
* margin of < 1cm between tumor edge and intestines
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 2 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 months
  Determination the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of carbon ion radiotherapy

SECONDARY OUTCOMES:
Progression-free Survival | Follow-up until progression up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

REFERENCES:
- [Derived] Hoegen-Sassmannshausen P, Naumann P, Hoffmeister-Wittmann P, Ben Harrabi S, Seidensaal K, Weykamp F, Mielke T, Ellerbrock M, Habermehl D, Springfeld C, Dill MT, Longerich T, Schirmacher P, Mehrabi A, Chang DH, Horner-Rieber J, Jakel O, Haberer T, Combs SE, Debus J, Herfarth K, Liermann J. Carbon ion radiotherapy of hepatocellular carcinoma provides excellent local control: The prospective phase I PROMETHEUS trial. JHEP Rep. 2024 Mar 11;6(6):101063. doi: 10.1016/j.jhepr.2024.101063. eCollection 2024 Jun. PMID 38737600
- [Derived] Habermehl D, Debus J, Ganten T, Ganten MK, Bauer J, Brecht IC, Brons S, Haberer T, Haertig M, Jakel O, Parodi K, Welzel T, Combs SE. Hypofractionated carbon ion therapy delivered with scanned ion beams for patients with hepatocellular carcinoma - feasibility and clinical response. Radiat Oncol. 2013 Mar 13;8:59. doi: 10.1186/1748-717X-8-59. PMID 23497349
- [Derived] Combs SE, Habermehl D, Ganten T, Schmidt J, Edler L, Burkholder I, Jakel O, Haberer T, Debus J. Phase i study evaluating the treatment of patients with hepatocellular carcinoma (HCC) with carbon ion radiotherapy: the PROMETHEUS-01 trial. BMC Cancer. 2011 Feb 12;11:67. doi: 10.1186/1471-2407-11-67. PMID 21314962